CLINICAL TRIAL: NCT03826251
Title: Nasogastric Tube After Small Bowel Obstruction Surgery is Not Mandatory: a Retrospective Cohort Study
Brief Title: Small Bowel Obstruction and Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: UH Angers 2018/75
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Acute Small Intestine Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- systematic nasogastric tube: NGT was left systematically after surgery and removed after the first flattus
- Non systematic nasogastric tube: Nasogastric tube was removed immediately after surgery and was replaced in case of vomiting
  Interventions: Procedure: Nasogastric tube removal

INTERVENTIONS:
Procedure: Nasogastric tube removal — Nasogastric tube was removed immediately after surgery
  Groups: Non systematic nasogastric tube

SUMMARY:
Postoperative management after small bowel obstruction (SBO) surgery is not consensual and better knowledge of risk factors for postoperative morbidity could help to add evidence of the feasibility of enhanced recovery programs (ERPs).

In elective surgery, ERPs have shown a significant benefit for the patient but this is not performed routinely in emergency surgery due to the difficulty to avoid postoperative nasogastric tube.

The aim was to identify risk factors for postoperative morbidity and for nasogastric tube (NGT) replacement after SBO surgery.

ELIGIBILITY:
Inclusion Criteria:

* Surgical management of Small bowel obstruction due to adhesions

Exclusion Criteria:

* obstruction not caused by single band adhesion
* matted adhesions, or if they were less than 18 years old

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgery for adhesive small bowel obstruction in the CHU of Angers between January 1, 2014 and December 31, 2017
Sampling Method: Probability Sample
Enrollment: 190
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
postoperative morbidity | within 30 days
  morbidity classified according to Dindo Clavien classification

SECONDARY OUTCOMES:
Nasogastric tube replacement | within 30 days
  nasogastric tube replacement after removal

IPD SHARING:
Plan to Share IPD: No